CLINICAL TRIAL: NCT04283760
Title: Investigation of the Reliability and Validity of the Movement Imagination Questionnaire - Revised Second in Acute Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatma Nurveren, Principal Investigator, Hacettepe University
Other Study IDs: GO 19/870
Record Dates: First submitted 2020-02-23; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Acute Stroke
Keywords: acute stroke; motor imagery; visual imagery; kinesthetic imagery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Group: 1. Demographic Information
  2. Mental Chronometry Test
  3. Movement Imagination Questionnaire- Revised Second
  4. Beck Depression Inventory
- Acute Stroke Patients: 1. Demographic Information
  2. Mental Chronometry Test
  3. Movement Imagination Questionnaire- Revised Second
  4. Beck Depression Inventory
  5. Trail Making Test
  6. Barthel Index
  7. Motor Assessment Scale
  8. Trunk Impairment Scale
  9. Mini Mental Test
  10. Glaskow Coma Scale

SUMMARY:
Our study was planned to investigate the reliability validity of the Movement Imagery Questionnaire- RS in acute stroke patients.

For our study, the Turkish version of the Movement Imagery Questionnaire-RS will be established first. Then, the reliability and validity of the questionnaire in acute stroke patients will be examined.

The study included 70 stroke patients hospitalized in the Stroke Unit of the Neurology Department of Hacettepe University Hospitals and individuals between 50-75 years of age who do not have any disease in Ankara.

DETAILED DESCRIPTION:
Motor imagery is a cognitive process that the person continues mentally without actually performing a particular motor movement. The concept of motor imaging has become more and more important in recent years and has allowed us to obtain different ideas about the emergence of motor movements. When the literature is analyzed, it was reported that the brain areas activated during the motor movement of individuals overlap with the active areas in the imaging process.As an individual's ability to imagine movement increases, the centers participating in the motor system become so activated. In the literature, it has been stated that this motor imaging ability may decrease in people who have had a stroke. For this reason, the motor imagination ability of the person should be evaluated before a suitable rehabilitation program is decided.When we look at the literature, it was seen that the Movement Imagery Questionnaire - Revised Second was used to evaluate the patients with subacute and chronic stroke, and there was no validity and reliability study in patients with acute stroke. Considering this situation, it was planned to translate the Movement Imagery Questionnaire -RS questionnaire into our language within the scope of our study and then to investigate the reliability and validity of patients with acute stroke.

ELIGIBILITY:
Inclusion Criteria:

Acute Stroke Patients:

* Ischemic stroke diagnosis by the relevant neurologist,
* At least 24 hours after stroke,
* Stroke for the first time
* Stable vital signs and no improvement in symptoms for 48 hours
* 50 to 75 years of age
* 15 points from Glaskow Coma Scale (GCS),
* Absence of apraxia and aphasia (apraxia and aphasia will be evaluated by the relevant neurologist.)
* Being able to walk at least 10 m independently
* A maximum score of 15 from the Beck Depression Inventory
* To score 24 or more from Mini Mental Test
* Signing the Informed Volunteer Consent Form

Healthy Group:

* Being in the 50-75 age range
* Signing the Informed Volunteer Consent Form
* A maximum score of 15 from the Beck Depression Inventory
* Not having a known neurological disease

Exclusion Criteria:

* Supplement for stroke patients; any neurological, orthopedic, psychological (such as schizophrenia, psychosis) and systemic problems for the healthy group
* Use of drugs to affect epilepsy, seizure attacks and cognition
* Cerebellum or mesencephalon lesion
* The presence of contractures or excessive spasticity in the joints to limit movement
* Neglect of a body half
* Irreversible visual (hemianopsia, blindness), presence of auditory disability
* Participate in another experimental or drug study during the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 70 stroke patients hospitalized in the Stroke Unit of the Neurology Department of Hacettepe University Hospitals and individuals aged 50-75 years living in Ankara who do not have any disease.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Movement Imagination Questionnaire - Revised Second | about 15 minutes
  Movement Imagination Questionnaire - Revised Second is a questionnaire used to evaluate motor imaging ability. The Movement Imagination Questionnaire has been revised especially for use in patients with motor function loss such as stroke. The questionnaire has 7 activities in total. Although most of these activities are sitting, there are also activities that must be done during standing. Each action is questioned both visually and kinesthetically and is scored based on the ease of visualization in the range of 0-7 points. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
The Motor Assessment Scale | about ten minutes
  The Motor Assessment Scale is designed to measure the functional properties of stroke patients. This assessment method evaluates the ability of stroke patients to perform functional tasks. The Motor Assessment Scale consists of eight motor tasks: (1) turning from the supine position, (2) sitting on your back, (3) sitting balance, (4) standing up, (5) walking, (6) upper limb function (7) hand gestures and (8) advanced hand gestures. In addition to these eight engines, the Motor Assessment Scale contains one more item that measures the overall tone. Each item is evaluated on a seven-degree scale from 0 to 6 (optimal motor behavior). The criterion for each degree in the scale corresponds to the description of the activity to be performed. In some cases, the maximum score (6 points) reflects the quality of performance; in others, it corresponds to performance over a period of time.
Mental Chronometry Test | about one minute
  Mental chronometry is an objective method used to evaluate motor imagery. It examines the time difference between actually making a movement and imagining the same movement. In general, in healthy individuals, the imagined movement time and movement time are related, but there are studies showing that this time is impaired in stroke patients. In our study, a 10 m walking test will be used to measure mental chronometry. First of all, the patient will be asked to walk 10 m independently and the time will be recorded. He will then be asked to imagine the movement and stop the stopwatch when he begins to imagine and stop himself again when he ends. Time difference and mental chronometry rate will be calculated.
Trail Making Test | about five minutes
  Trail Making Test It is used to evaluate individuals' visual scanning speed, managerial functions, visual-motor perception, motor function, planning, organization, abstract thinking and response limitation. The test consists of 2 parts, A and B. In section A, the individual is asked to combine the numbers from 1 to 25 and completion time is recorded. In section B, the individual completes the ordering, corresponding to a number and a letter, respectively, and the completion time is recorded.
Barthel Index | about 5 minutes
  Barthel Index evaluates the basic activities of daily life in order to determine at what level individuals can independently determine activities such as nutrition, washing, self-care, dressing, bowel care and bladder care, sitting on the toilet, going from bed to wheelchair, using walking / wheelchair and climbing stairs. It is a 10-item scale. The scale has scoring ranging from 0 to 20 or 0 to 100 depending on the daily life activities.
Mental Chronometry Ratio | about one minute
  Real performance time - imagery time/ real performance time
Trunk Impairment Scale | about one minute
  Trunk Impairment Scale is a scale that evaluates post-stroke body disorder. The scale, consisting of 7 parameters, also includes perception of vertical posture, trunk rotation muscle strength and reflexes on the affected and unaffected side, and vertical stop and abdominal manual muscle test sub parameters in Tsuji and colleagues' stroke disorder evaluation set. Each parameter is evaluated over 4 points. The total score ranges from a minimum of 0 to a maximum of 21 points. A higher score means better performance. In this study, only the vertical stop subscale of this scale will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Üniversitesi, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Butler AJ, Cazeaux J, Fidler A, Jansen J, Lefkove N, Gregg M, Hall C, Easley KA, Shenvi N, Wolf SL. The Movement Imagery Questionnaire-Revised, Second Edition (MIQ-RS) Is a Reliable and Valid Tool for Evaluating Motor Imagery in Stroke Populations. Evid Based Complement Alternat Med. 2012;2012:497289. doi: 10.1155/2012/497289. Epub 2012 Feb 28. PMID 22474504
- [Background] Gregg M, Hall C, Butler A. The MIQ-RS: A Suitable Option for Examining Movement Imagery Ability. Evid Based Complement Alternat Med. 2010 Jun;7(2):249-57. doi: 10.1093/ecam/nem170. Epub 2007 Dec 26. PMID 18955294
- [Background] Greiner J, Schoenfeld MA, Liepert J. Assessment of mental chronometry (MC) in healthy subjects. Arch Gerontol Geriatr. 2014 Mar-Apr;58(2):226-30. doi: 10.1016/j.archger.2013.09.003. Epub 2013 Oct 18. PMID 24275122
- [Background] Malouin F, Pichard L, Bonneau C, Durand A, Corriveau D. Evaluating motor recovery early after stroke: comparison of the Fugl-Meyer Assessment and the Motor Assessment Scale. Arch Phys Med Rehabil. 1994 Nov;75(11):1206-12. doi: 10.1016/0003-9993(94)90006-x. PMID 7979930
- [Background] Cangoz B, Karakoc E, Selekler K. Trail Making Test: normative data for Turkish elderly population by age, sex and education. J Neurol Sci. 2009 Aug 15;283(1-2):73-8. doi: 10.1016/j.jns.2009.02.313. Epub 2009 Mar 4. PMID 19264326
- [Background] Tsuji T, Liu M, Sonoda S, Domen K, Chino N. The stroke impairment assessment set: its internal consistency and predictive validity. Arch Phys Med Rehabil. 2000 Jul;81(7):863-8. doi: 10.1053/apmr.2000.6275. PMID 10895996
- [Background] Fujiwara T, Liu M, Tsuji T, Sonoda S, Mizuno K, Akaboshi K, Hase K, Masakado Y, Chino N. Development of a new measure to assess trunk impairment after stroke (trunk impairment scale): its psychometric properties. Am J Phys Med Rehabil. 2004 Sep;83(9):681-8. doi: 10.1097/01.phm.0000137308.10562.20. PMID 15314532
- [Background] Fu C, Jin X, Chen B, Xue F, Niu H, Guo R, Chen Z, Zheng H, Wang L, Zhang Y. Comparison of the Mini-Mental State Examination and Montreal Cognitive Assessment executive subtests in detecting post-stroke cognitive impairment. Geriatr Gerontol Int. 2017 Dec;17(12):2329-2335. doi: 10.1111/ggi.13069. Epub 2017 Jul 4. PMID 28675607